CLINICAL TRIAL: NCT06292208
Title: Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetic (PK) and Preliminary Efficacy of IBD0333 in Patients With Locally Advanced/Metastatic Solid Tumor or Non-Hodgkin Lymphoma
Brief Title: A Clinical Trial to Evaluate Effect of IBD0333 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBD0333-101
Record Dates: First submitted 2024-01-31; First posted 2024-03-05 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: MTD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IBD0333 (Experimental)
  Interventions: Biological: IBD0333

INTERVENTIONS:
Biological: IBD0333 — This is a phase I/II, open, non-randomized, dose-escalation and expansion study designed to evaluate the safety, tolerability, pharmacokinetic (PK), immunogenicity, and preliminary efficacy of IBD0333 in patients with locally advanced/metastatic solid tumor or non-Hodgkin lymphoma in dose-escalation, dose-expansion, and clinical exploration phases.

SUMMARY:
Primary Objectives Dose escalation phase To evaluate the safety and tolerability of IBD0333 in patients with locally advanced/metastatic solid tumor or non-Hodgkin lymphoma and to determine the maximum tolerated dose (MTD), extended recommended dose (DRDE), and/or dose limiting toxicity (DLT).

Dose expansion phase To evaluate the safety and tolerability of IBD0333 in patients with locally advanced/metastatic solid tumor or non-Hodgkin lymphoma and to determine the recommended Phase 2 dose (RP2D).

Clinical exploration phase To evaluate the preliminary efficacy of IBD0333 in patients with specific tumor.

Secondary objectives Dose escalation phase & Dose expansion phase To evaluate the pharmacokinetic (PK) of IBD0333 in patients with locally advanced/metastatic solid tumor or non-Hodgkin lymphoma; To evaluate the immunogenicity of IBD0333 in patients with locally advanced/metastatic solid tumor or non-Hodgkin lymphoma; To evaluate the preliminary efficacy of IBD0333 in patients with locally advanced/metastatic solid tumor or non-Hodgkin lymphoma.

Clinical exploration Phase To evaluate the safety and tolerability of IBD0333 in patients with specific tumor; To evaluate the immunogenicity of IBD0333 in patients with specific tumor. Exploratory Objectives To explore biomarkers in blood and tissue that predict potential efficacy of IBD0333.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible for participation in this trial, the patient must:

1. Male or female, 18 to 80 years old.
2. Patients with histologically or cytologically confirmed locally advanced/metastatic solid tumor or non-Hodgkin lymphoma who have failed or have no standard therapy, or for whom the standard therapy is intolerant.
3. There is at least one assessable tumor lesion in the dose escalation phase and at least one measurable lesion in the dose expansion phase according to RECIST 1.1 (solid tumors) or Lugano 2014 (lymphomas) (tumor lesions located in areas of prior radiotherapy or other localized regional treatment areas are generally not considered as measurable lesions unless the lesion shows definite progression or persists after 3 months of radiotherapy).
4. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
5. Have a life expectancy of at least 3 months.
6. Have adequate organ function as indicated by the following laboratory values.

   1. Hematological (no transfusion or hematopoietic stimulating factor therapy within 14 days): absolute neutrophil count (ANC)≥1.5×109/L, platelet count (PLT)≥ 90 ×109/L, hemoglobin (HGB)≥90 g/L;
   2. Hepatic: total bilirubin (TBIL)≤1.5×upper limit of normal (ULN), except for Gilbert syndrome; alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤3.0×ULN, or ALT and AST ≤ 5.0×ULN in patients with liver metastases or liver cancer;
   3. Renal: creatinine clearance (Ccr)≥50mL/min (calculated according to the Cockcroft-Gault Method:);
   4. Coagulation: international normalized ratio (INR) ≤ 1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN.
7. Eligible patients (male and female) of childbearing potential must agree to use a reliable contraception measure (hormonal or barrier contraception or abstinence) with their partner for the duration of the trial and for at least 120 days after the discontinuation of investigational product. Female patients of childbearing potential must have a negative serum pregnancy test at within 7 days of first dose of investigational product.
8. According to the investigator's assessment, the patient could benefit from IBD0333.
9. Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment.

Exclusion Criteria

1. Known hypersensitivity reaction (NCI-CTCAE 5.0 ≥ grade 3) recombinant proteins or any excipient contained in the drug or vehicle formulation for IBD0333.
2. History of 4-1BB monoclonal antibody or 4-1BB-containing dual antibody immune costimulatory molecule agonist.
3. History of anti-cancer therapies prior to the initiation of investigational product (chemotherapy within 3 weeks; radiotherapy, biologic therapy, endocrine therapy, targeted therapy, immunotherapy within 4 weeks) and the following are except:

   1. Nitrosourea or mitomycin C within 6 weeks prior to the initiation of investigational product;
   2. Oral fluorouracil and small molecule-targeted drugs within 2 weeks prior to the initiation of investigational product;
   3. Chinese patent drugs within 2 weeks prior to the initiation of investigational product.
4. History of investigational anti-cancer drug within 4 weeks prior to the initiation of investigational product.
5. History of major surgery (except for puncture biopsy) or significant trauma within 4 weeks prior to the initiation of investigational product, or require the selective surgery during the trial.
6. History of systemic corticosteroids (prednisone >10 mg/day or equivalent) or immunosuppressive medication <14 days prior to the initiation of investigational product. Steroids for topical, ocular, intra-articular, intranasal and inhaled and short-term prophylactic treatment (e.g., to prevent contrast allergy) were allowed.
7. Treatment with immunomodulatory agents within 14 days prior to the initiation of investigational product, including but not limited to thymidine, interleukin-2, interferon, etc.
8. Vaccination with live attenuated vaccine within 4 weeks prior to the initiation of investigational product.
9. History of allogeneic hematopoietic stem cell or organ transplantation.
10. The adverse effects related to prior anticancer treatment (except alopecia, peripheral neurotoxicity with grade 2, and stable hypothyroidism after hormone replacement therapy or the other toxicities judged by the investigator without safety risk) that have not resolved to ≤ Grade 1 according to common terminology criteria for adverse events (NCI-CTCAE 5.0) or relevant provisions of the inclusion criteria prior to initiation of investigational product.
11. Parenchymal brain metastases or meningeal metastases unless previously received therapies and have no evidence of progression on magnetic resonance imaging (MRI) or computed tomography (CT) for at least 8 weeks after the treatment and for 4 weeks prior to the initiation of investigational product.
12. Evidence of active infection requiring intravenous systemic therapy.
13. History of immunodeficiency, including the positive for human immunodeficiency virus (HIV) antibodies.
14. Active hepatitis B infection (HBsAg positive and HBV-DNA > 500 IU/mL or lower limit of detection [only if lower limit is above 500 IU/mL]). Active hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
15. Has interstitial lung disease (except for the radiographic pulmonary fibrosis without hormone therapy).
16. History of serious cardiovascular disease, including but not limited to:

    1. Have severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III-degree atrioventricular block, etc.;
    2. The mean QT interval corrected for heart rate by Fridericia's formula (QTcF) >470msec.
    3. History of acute coronary syndromes, congestive heart failure, aortic dissection, stroke or other cardiovascular or cerebrovascular ≥ grade 3 within the 6 months prior to initiation of investigational product.
    4. Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system or left ventricular ejection fraction (LVEF) < 50%, or structural heart disease with high risk judged by investigators;
    5. Uncontrollable hypertension.
17. Previous or current autoimmune disease (systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for the stable autoimmune thyroid disease, type I diabetes, vitiligo, cured atopic dermatitis in children, and psoriasis (within the past 2 years and without systemic therapy).
18. History of ≥Grade 3 Immune-Related Adverse Events (irAE) or ≥Grade 2 immune-associated myocarditis (experienced immune-associated thyroid toxicity ≥grade 3 could be enrolled).
19. History of malignancy or current other malignant tumors (other than in non-melanoma skin cancer, localized prostate cancer, carcinoma in situ [situ cervical cancer] treated with curative intent and without evidence of disease for 2 years or longer).
20. Has uncontrollable third interstitial fluid that are unsuitable for enrollment (judged by the investigator).
21. Has alcohol or drug dependence.
22. Has a psychiatric disorder or poor compliance.
23. Pregnant or breastfeeding. Have serious systemic disease or are unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD | through study completion, an average of 1 year
  Maximum tolerated dose
DRDE | through study completion, an average of 1 year
  Extended recommended dose
Dose limiting toxicity (DLT) | 28 days after first dose(dose-escalation phase)
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
RP2D | through study completion, an average of 1 year
  Recommended Phase 2 dose
ORR | through study completion, an average of 1 year
  Objective response rate

SECONDARY OUTCOMES:
pharmacokinetic parameters | through study completion, an average of 1 year
  AUC0-t
pharmacokinetic parameters | through study completion, an average of 1 year
  Cmax
pharmacokinetic parameters | through study completion, an average of 1 year
  Tmax
pharmacokinetic parameters | through study completion, an average of 1 year
  t1/2
ADA | through study completion, an average of 1 year
  Anti-drug antibody
ORR | through study completion, an average of 1 year
  Objective response rate
DCR | through study completion, an average of 1 year
  Disease control rate
DoR | through study completion, an average of 1 year
  Duration of relief
PFS | through study completion, an average of 1 year
  Progression-free survival
Frequency of adverse events (AEs) and SAEs | through study completion, an average of 1 year
  To investigate the safety characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided